CLINICAL TRIAL: NCT05620420
Title: A Multicenter Cross-sectional Study on Mental Health of Patients With Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2022-068-A
Record Dates: First submitted 2022-11-10; First posted 2022-11-17 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Psychological Distress; Insomnia; Somatic Symptoms
Keywords: multiple myeloma; mental health
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Medically Unexplained Symptoms; Multiple Myeloma; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multiple myeloma patients with normal ability of communication and understanding will be enrolled. DT, GAD-7, PHQ-15 and PSQI scales are designed to assess the mental health status of the patients. Demographic and disease data of patients will be collected as well. The main aim is to explore the factors affecting the mental health of myeloma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic multiple myeloma were diagnosed according to the criteria of Chinese multiple myeloma diagnosis and treatment guidelines (revised in 2022).
2. Age ≥18 years, with junior high school education or above. Patients have normal ability of communication and understanding.
3. Informed consent has been signed.

Exclusion Criteria:

1. Who has kinship with other enrolled patients.
2. Life expectancy of< 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited form 14 medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
morbidity of psychological distress in patients with multiple myeloma. | Baseline (the time when the patient is enrolled to the study)
  The total score of DT scale ≥4 points is defined as obviously psychological distress.

SECONDARY OUTCOMES:
morbidity of anxiety in patients with multiple myeloma. | Baseline (the time when the patient is enrolled to the study)
  GAD-7 scale is applied to assess the anxiety of the patient
morbidity of insomnia in patients with multiple myeloma. | Baseline (the time when the patient is enrolled to the study)
  PSQI scale is applied to assess the insomnia of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Jian Hou, Principal Investigator — RenJi Hospital
Locations (1):
- shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality, China